CLINICAL TRIAL: NCT02569879
Title: Impact of Boostrix™ Maternal Vaccination on Morbidity and Mortality of Pertussis Disease in Infants ≤6 Weeks of Age, in Bogota, Colombia.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201521
Record Dates: First submitted 2015-10-01; First posted 2015-10-07 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diphtheria; Acellular Pertussis; Tetanus; Aspergillosis, Allergic Bronchopulmonary; Diphtheria-Tetanus-acellular Pertussis Vaccines
Keywords: Boostrix™; Bagota; maternal vaccination; Pertussis; Mortality; Morbidity
MeSH Terms: conditions — Diphtheria; Tetanus; Aspergillosis, Allergic Bronchopulmonary; Whooping Cough

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Infants Group: * All infants ≤12 months of age in Bogota, reported with pertussis disease in the national databases of Bogota, between January 2005 and December 2014.
  * All infants ≤12 months of age in Bogota, deceased between January 2005 and December 2014 due to pertussis disease (primary diagnosis), based on death certificate information.
  * All infants ≤12 months of age in Bogota, with ALRTI, between January 2005 and December 2014.
  * All infants ≤12 months who have received primary pertussis vaccination in Bogota, between January 2005 and December 2014.
  Interventions: Other: Pertussis maternal immunization
- Pregnant women Group: • Pregnant women will be included in the study to assess the vaccination coverage of Boostrix from March 2013 to December 2014
  Interventions: Other: Pertussis maternal immunization

INTERVENTIONS:
Other: Pertussis maternal immunization — Retrospective time trend analysis before and after pertussis maternal immunization in Bogota, Colombia.

SUMMARY:
This study is being conducted to assess impact of maternal immunisation against pertussis in infants ≤12 months of age before and after introduction of pertussis maternal immunisation in Bogota, Colombia from January 2005-December 2014.

DETAILED DESCRIPTION:
An observational, retrospective, ecological database study which involves systematic screening of the national databases of Bogota, to study pertussis related morbidity and mortality in infants ≤ 12 months of age before and after introduction of pertussis maternal immunisation in Bogota, Colombia from January 2005-December 2014.

ELIGIBILITY:
Inclusion Criteria:

• Not applicable as since this retrospective database study will include all the available aggregated data of pertussis cases, pertussis related hospitalisations and deaths, ALRTI cases, primary pertussis vaccination coverage and Boostrix vaccination coverage.

Exclusion Criteria:

• Not applicable as since this retrospective database study will include all the available aggregated data of pertussis cases, pertussis related hospitalisations and deaths, ALRTI cases, primary pertussis vaccination coverage and Boostrix vaccination coverage.

Ages: 0 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: * All infants ≤12 months of age in Bogota, reported with pertussis disease in the national databases of Bogota, between January 2005 and December 2014.
  * All infants ≤12 months of age in Bogota, deceased between January 2005 and December 2014 due to pertussis disease (primary diagnosis), based on death certificate information.
  * All infants ≤12 months of age in Bogota, with ALRTI, between January 2005 and December 2014.
  * All infants ≤12 months who have received primary pertussis vaccination in Bogota, between January 2005 and December 2014.
  * All pregnant women who have received Boostrix as a part of the UMV program in Bogota, between March 2013 and December 2014.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-04-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of reported cases of hospitalisations and deaths due to pertussis in infants ≤6 weeks of age, in post-vaccination period compared to pre-vaccination period of Boostrix vaccination | During the 9-year period (January 2005- December 2014)

SECONDARY OUTCOMES:
Occurrence of reported cases of hospitalisations and deaths due to pertussis in infants 7 weeks to ≤12 months of age, in post-vaccination period compared to pre-vaccination period of Boostrix vaccination | During the 9-year period (January 2005- December 2014)
Occurrence of ALRTI in infants ≤6 weeks of age and 7 weeks to ≤12 months of age, following the introduction of pertussis maternal immunisation in Bogota, Colombia | During the 9-year period (January 2005- December 2014)
Description of the total number of doses of Boostrix administered in pregnant women, after its introduction into the UMV program in Bogota | During the 9-year period (January 2005- December 2014)
Description of the total number of doses of primary pertussis vaccine administered to infants ≤12 months of age in Bogota | During the 9-year period (January 2005- December 2014)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrasquilla G, Porras A, Martinez S, DeAntonio R, Devadiga R, Caceres DC, Juliao P. Incidence and mortality of pertussis disease in infants <12 months of age following introduction of pertussis maternal universal mass vaccination in Bogota, Colombia. Vaccine. 2020 Oct 27;38(46):7384-7392. doi: 10.1016/j.vaccine.2020.07.046. Epub 2020 Oct 2. PMID 33012607